CLINICAL TRIAL: NCT03189056
Title: Lower Urinary Tract Dysfunction in Chronic Chagas' Disease : Clinical and Urodynamic Presentation
Status: Completed | Type: Observational
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Elsa BEY, Resident in urological surgery, Institut de Recherche pour le Developpement
Other Study IDs: Chagas_urology
Record Dates: First submitted 2017-06-09; First posted 2017-06-16 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Chagas' Disease (Chronic) With Other Organ Involvement
Keywords: chronic Chagas disease; bladder; lower urinary tract; urodynamic
MeSH Terms: conditions — Chagas Disease; Bronchiolitis Obliterans Syndrome | interventions — Creatinine

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single cohort: single cohort for transversal study patients presenting chronic chagas disease for all patients : clinical examination/questionnaires/ quality of life/ blood sample for renal function (creatinina) and Chagas serology control if needed/ uroflowmetry/ ultrasonography
  If symptomatic patient at first exploration : urodynamic exploration is proposed (cystomanometry, urethral profile, pressure/flow study). No electromyograma. No video urodynamic procedure.
  Interventions: Diagnostic Test: Chagas serology; Biological: Creatinina; Procedure: Urodynamic exploration

INTERVENTIONS:
Diagnostic Test: Chagas serology — IFI + ELISA method if no biological confirmation of chagas disease is in our possession
Biological: Creatinina — Plasmatic single mesure after consultation 1, to evaluate renal function
Procedure: Urodynamic exploration — With a new equipement SmartDyn Albynmedical imported from Spain for the study Single use sterile equipment shipped Control of urine sterility before procedure Informed consent signed If acquired urinary infection after procedure, patient treated free of charge and clinical evolution controlled

SUMMARY:
Chagas disease is one of the most neglected vector-borne infectious disease worldwide. The first decades following the discovery of the pathology drove an international research enthusiasm, mainly concentrated on understanding the typical cardiac and digestive forms. Recently, research have been focused on vector control, which has been a huge success, at the price of neglecting the patients who already presented fixed and severe organic lesions due the chronic phase of the illness.

This study focus on a rarely studied aspect of this pathology: the involvement of the lower urinary tract and it's symptomatology in adults suffering from Chagas chronic disease.

Various studies have assessed the involvement of the lower urinary tract in chronic Chagas disease, the vast majority of them being on the animal model or very ancient human studies mainly on cadaveric specimen, the first of them being the primary description of Koeberle in 1963.

Human symptomatology deriving from bladder, ureteral and urethral chronic chagasic lesions are yet widely unknown, and only a few Brazilian and Mexican studies have intended to describe the clinical and urodynamic presentation of these patients.

The aim of this study is to assess the prevalence of urinary disorders in chronic chagasic patients and to describe their symptoms, through a complete clinical, ultrasonographic and urodynamic description.

DETAILED DESCRIPTION:
Epidemiologic observationnal transversal study

Cohort of patients between 18 and 50 years of age, presenting a chronic form of Chagas' disease (cardiopathy, mega-colon or mega-esofagus), and presenting non of the exclusion criteria.

Recruitment via the existing patients list of positive Chagas serology of:

* the SELADIS center (Instituto de Servicios de Laboratorio de Diagnostico e Investigacion en Salud UMSA -UNIVERSIDAD MAYOR DE SAN ANDRES-)
* Private surrounding hospitals, Hospital de Clinicas and Centro de Seguro Social Universitario de La Paz (UMSA)
* Laboratorio de Inmunodiagnostico Instituto Boliviano de Biologia de la Altura -IBBA-Dr Lourdes Echalar.

Informed consent signed.

1 to 3 consultations on a period of one to 2 weeks no follow-up (transversal study)

Invasive descriptive explorations (blood sample and urodynamic study, imposing the assent of the Comité Nacional de Bioética).

Main objective : Describe the prevalence of the lower urinary tract dysfunction in patients suffering from a chronic form of Chagas' disease. The main criteria evaluated is the sum of two symptom questionnaires IPSS and ICIQ (spanish official validated translation), focusing on urinary incontinence, voiding dysfunction and quality of life.

Secondary objectives :

All the included patients will be proposed an initial consult :

* Anonymization of all the observation/results
* Past history (pathology, actual treatment,…), search of the exclusion criteria, Chagas' disease symptomatology and treatment, urological symptomatology.
* Validated questionnaires to evaluate urological symptoms, urinary incontinence, voiding dysfunction or acute urinary dysfunction, bladder hyperactivity, sexuality and fertility.
* Clinical examination
* Micturition calendar /48hours.
* Uroflowmetry, followed by ultrasonography for post-void residual and upper-urinary tract dilatation.
* Blood sample to evaluate renal function (plasmatic creatinina for CDK EPI formula). This blood sample can also be used to confirm the positive Chagas' serology if no serology is available (indirect immunofluorescence and ELISA).

Te participants presenting a symptomatic lower urinary tract dysfunction on the previous exams will be proposed a complete urodynamic exploration (cystomanometry, urethral profile, pression/flow study during mycturition).

Sterility of urine assessed before exam. Tecnical material imported from Spain, Albyn medical Smardyn and consummables. Electronic curves obtained from Phoenix software (Albyn).

Objective inclusion of 200 participants during 5 months, between June and October 2017, in the SELADIS Institute in La Paz, Bolivia. Director of study Dr Simone Frédérique Brenière (french), Bolivian Director of Institute Dra Susana Revollo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 50 years of age
* Presenting a chronic form of Chagas disease : cardiopathy or enteropathy
* Previously treated or not treated
* Signed informed consent

Exclusion Criteria:

* Diabetes
* Neurologic pathology
* Past history of extensive pelvic surgery
* Vaginal prolaps > grade 3 of Baden & Walker (female)
* Past history of vertebral fracture > L2

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients presenting a chronic form of chagas disease diagnosed by the SELADIS institute (serology), by cardiology, gastro-enterology or infectious disease consultation in La Paz may be include, after the informed consent have been signed.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2017-10-20 (Actual); Study Completion 2017-10-20 (Actual)

PRIMARY OUTCOMES:
Symptomatic patients | at consultation : 1 day (transversal study, the participant will not be followed)
  ICIQ SF>0 IPSS>7 or past acute urinary retention IIEF5<11

SECONDARY OUTCOMES:
Megabladder | at consultation : 1 day (transversal study, the participant will not be followed)
  Bladder capacity >600cc and <4 daily micturition
Mega ureter | at consultation : 1 day (transversal study, the participant will not be followed)
  Ultrasonographic dilatation of renal pelvis>20mm or of ureter >7mm
Hyperactive bladder | micturition calendar over 2 days (transversal study, the participant will not be followed)
  >8 daily micturition + urgency on dairy subsection detrusor hyperactivity on cystomanometry
Detrusor underactivity | at consultation : 1 day (transversal study, the participant will not be followed)
  Qmax<15 mL/s and post void residual>150cc per-micturition pressure <40 cm H2O
Renal insufficiency | at consultation : 1 day (transversal study, the participant will not be followed)
  CDK EPI<60 mL/mn
Urinary recurrent infections | reported infections duing the last 5 years (transversal study, the participant will not be followed)
  past history > 3 pyélonephritis or >5 cystitis/year in the past 5 years, if associated with dilatated ureter/renal pelvis or significant post void residual
Urinary sphincter insufficiency | at consultation : 1 day (transversal study, the participant will not be followed)
  P max<30 cm H20 and stress urinary incontinence
Erectile dysfunction in males | at consultation : 1 day (transversal study, the participant will not be followed)
  IIEF5 <16
Hypofertility | at consultation : 1 day (transversal study, the participant will not be followed)
  oral assess by difficulty to obtain pregnancy >1 year

CONTACTS AND LOCATIONS:
Overall Officials: Elsa BEY, Resident, Principal Investigator — IRD
Locations (1):
- SELADIS Institute, Universidad Mayor de San Andrès, La Paz, Bolivia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Jelicks, Linda A., et Herbert B. Tanowitz. " Advances in Imaging of Animal Models of Chagas Disease ". Advances in Parasitology 75 (2011): 193-208. doi:10.1016/B978-0-12-385863-4.00009-5. — https://doi.org/10.1016/B978-0-12-385863-4.00009-5
- See also: Ny, Lars et al. " A Magnetic Resonance Imaging Study of Intestinal Dilation in Trypanosoma Cruzi-Infected Mice Deficient in Nitric Oxide Synthase ". The American Jour — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC2701742/
- See also: Ardito et al. " Chronic Renal Impairment in Patients with Chagas Cardiomyopathy with Chronic Systolic Heart Failure: Prevalence and Prognostic Significance ". Inte — http://dx.doi.org/10.1016/j.ijcard.2011.07.060
- See also: Koeberle, F. " ENTEROMEGALY AND CARDIOMEGALY IN CHAGAS DISEASE ". Gut 4 (décembre 1963): 399-405. — https://www.ncbi.nlm.nih.gov/pubmed/14084752
- See also: Mirkin et al. " Experimental Chagas' Disease: Electrophysiology and Cell Composition of the Neuromyopathic Inflammatory Lesions in Mice Infected with a Myotropic and a Pantropic Strain of — https://www.ncbi.nlm.nih.gov/pubmed/9030871
- See also: Cabrine-Santos et al. " Genitourinary Changes in Hamsters Infected and Reinfected with Trypanosoma Cruzi ". Memórias Do Insti — https://www.ncbi.nlm.nih.gov/pubmed/12937767
- See also: Scremin, L. H., C. E. Corbett, M. D. Laurenti, E. V. Nunes, J. J. Gama-Rodrigues, et M. Okumura. " Megabladder in Experimental Chagas Disease: Pathological Features of the Bladder Wall ". Revista Do Hospital Das Clínicas 54, nᵒ 2 (avril 1999): 43-46. — https://www.ncbi.nlm.nih.gov/pubmed/10513065
- See also: Suaid et al. " Modulation of Urethral Alpha-Sympathetic by Parasympathetic before and Following Bethanechol Chloride Injection ". International Braz J Urol: Official J — https://www.ncbi.nlm.nih.gov/pubmed/15745502
- See also: DeFaria, C. R., J. M. De Rezende, et A. Rassi. " [Peripheral denervation in the various clinical forms of Chagas' disease] ". Arquivos De Neuro-Psiquiatria 46, nᵒ 3 (septembre 1988): 225-37. — https://www.ncbi.nlm.nih.gov/pubmed/2851967
- See also: Carraro, A. A., R. A. Lopes, R. D. Ribeiro, et T. L. Lamano Carvalho. " The Male Reproductive Organs in the Chronic Phase of Experimental Chagas' Disease ". Angewandte Parasitologie 33, nᵒ 1 (février 1992): 3-9. — https://www.ncbi.nlm.nih.gov/pubmed/1590593
- See also: Rocha, J. N., H. J. Suaid, A. C. P. Martins, A. J. Cologna, S. Tucci Jr., et M. A. Gonçalves. " URODYNAMIC ASSESSEMENT IN PATIENTS WITH CHAGAS DISEASE ". Acta Cirurgica Brasileira 16 (2001): 7-8. doi:10.1590/S0102-86502001000500003. — http://www.scielo.br/scielo.php?script=sci_abstract&pid=S0102-86502001000500003&lng=en&nrm=iso&tlng=pt